CLINICAL TRIAL: NCT02146508
Title: Endoscopic Prevention of Esophageal Cancer at Tenwek Hospital (The EXPECT Trial) by Removal or Ablation of Esophageal Squamous Cell Dysplasia
Brief Title: Endoscopic Prevention of Esophageal Cancer at Tenwek Hospital
Acronym: EXPECT
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Medtronic owns Covidien & closed study 11/18/15. Will reapply through Medtronic.
Sponsor: Tenwek Hospital (Other)
Collaborators: Mayo Clinic (Other); National Cancer Institute (NCI) (NIH); Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Stephen Burgert, Director of Endoscopy Services, Tenwek Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P62/02/2013
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Esophageal Cancer; Esophageal Squamous Dysplasia
Keywords: Esophageal cancer; Radiofrequency, catheter ablation; Endoscopic mucosal resection; Esophageal squamous dysplasia; Cancer prevention
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Endoscopic Mucosal Resection; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic treatment (Experimental): Participants undergo upper GI endoscopy with endoscopic mucosal resection (EMR) and/or radiofrequency ablation (RFA) of esophageal squamous dysplasia (ESD). After initial therapy participants undergo repeat endoscopy every 3 months for a year, with re-biopsy and re-treatment of residual ESD as appropriate.
  Interventions: Procedure: Endoscopic Mucosal Resection (EMR); Device: Radiofrequency ablation

INTERVENTIONS:
Procedure: Endoscopic Mucosal Resection (EMR) — Endoscopic removal of regions of ESD.
Device: Radiofrequency ablation — Endoscopic radiofrequency ablation of regions of ESD
  Other Names: HALO360 (Covidien, Inc.); HALO90 (Covidien, Inc.); HALO60 (Covidien, Inc.)

SUMMARY:
Esophageal cancer is common in Kenya. The precursor of esophageal cancer is esophageal squamous dysplasia (ESD). In this study, persons known to have ESD will undergo endoscopic removal or ablation of ESD in order to prevent development of esophageal cancer.

DETAILED DESCRIPTION:
Esophageal squamous dysplasia (ESD) is the precursor lesion of esophageal squamous cell cancer. ESD causes no symptoms but can be detected by screening. ESD may harbor various grades of dysplasia. Patients with moderate grade or high grade dysplasia (MGD or HGD) have up to a 40-fold increased risk of esophageal squamous cell cancer.

In this study, persons known to have ESD with MGD or HGD on the basis of prior screening will be invited to undergo endoscopic treatment with either endoscopic mucosal resection (EMR) and/or radio frequency ablation (RFA) in order to remove or ablate regions of ESD. Participants will undergo a series of endoscopies to treat ESD and monitor success of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant is 18-85 years of age, inclusive
* Participant has had a prior endoscopy with Lugol's chromoendoscopy demonstrating an unstained lesion (USL) of at least 5 mm which on biopsy contained moderate grade dysplasia (MGD), high grade dysplasia (HGD), or esophageal squamous cell cancer (ESCC) of flat mucosa limited to the lamina propria, with no evidence of invasion.
* The maximum allowable linear length of USL-bearing esophagus is 20 cm.
* No more than 14 continuous linear cm of esophagus require treatment for MGD, HGD, or ESCC.
* For patients with ESCC, CT scan of chest and upper third of the abdomen shows no exclusionary findings for the trial, such as metastasis.
* Participant is not pregnant and has no plans to become pregnant in the ensuing 12 months (confirmation of pregnancy status in women of child-bearing age and ability required prior to each endoscopy with urine or blood test, if subject believes she may be pregnant or has missed a menstrual period)
* Participant is eligible for treatment and follow-up endoscopy and biopsy as required by the protocol
* Participant is willing to provide written, informed consent to participate in this clinical study and understands the responsibilities of trial participation

Exclusion Criteria:

* Esophageal stricture preventing passage of a therapeutic endoscope
* Any prior endoscopic resection
* Any esophageal dilation in the past 12 months
* Any history of ESCC of the esophagus, except for ESCC of flat mucosa limited to the lamina propria diagnosed within 12 months of study enrollment.
* In participants with ESCC, any evidence of nodal involvement or distant metastases
* Any previous ablative therapy within the esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, laser treatment, or other) or any radiation therapy to the esophagus.
* Any previous esophageal surgery, except fundoplication
* Evidence of esophageal varices detected within last 6 months or at initial EMR/RFA procedure
* Evidence of eosinophilic esophagitis on endoscopy and/or histology
* History of coagulopathy, or use of warfarin within the past month.
* Report of uncontrolled coagulopathy with international normalized ratio (INR) > 2 or platelet count <75,000 platelets per µL (note: laboratory testing is not required for all subjects in this study)
* Participant is using aspirin, clopidogrel, or non-steroidal anti-inflammatory drugs that cannot be discontinued 7 days before and after therapeutic sessions
* Participant has a known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines
* Participant has an implantable pacing device (examples; automatic implantable cardioverter/defibrillator, neurostimulator, cardiac pacemaker) and has not received clearance for enrollment in this study by the physician responsible for the pacing device
* Participant suffers from psychiatric or other illness deemed by the investigator as an inability to comply with protocol
* Participant has life expectancy less than 2 years

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2013-06; Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Complete resolution of advanced esophageal squamous dysplasia | 12 months
  The percentage of subjects demonstrating complete response defined as complete histological clearance of MGD, HGD and esophageal squamous carcinoma in the treatment areas at 12 months after the initial ablation procedure.

SECONDARY OUTCOMES:
Safety of endoscopic interventions | 12 months
  Percentage of participants experiencing serious adverse events following EMR or RFA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Burgert, MD, Principal Investigator — Tenwek Hospital
Locations (1):
- Tenwek Hospital, Bomet, Kenya